CLINICAL TRIAL: NCT01884701
Title: Accessing Peripheral Occluded LesiOns II (APOLO-II)
Acronym: APOLO-II
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCross Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVO-031
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2015-03

CONDITIONS: Femoropopliteal Occlusive Disease
Keywords: Chronic Total Occlusion CTO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Intervention
  Interventions: Device: ENABLER-P Catheter System

INTERVENTIONS:
Device: ENABLER-P Catheter System

SUMMARY:
The current study is a prospective, single-arm, non-randomized, multi-center study to evaluate the outcome of the ENABLER-P Catheter System for crossing chronic total occlusions during endovascular intervention for femoral-popliteal occlusive disease.

ELIGIBILITY:
Inclusion Criteria:

* Documentation from a previous attempt OR a concurrent reasonable attempt (at least 5 minutes) during this procedure, demonstrating resistance to conventional guidewire crossing;
* Patient must have objective evidence of lower extremity ischemia;
* Totally occlusive lesion in a native femoropopliteal artery classified angiographically as absolute (100% occlusion with no flow), where no antegrade filling beyond the occlusion is visible;
* Target occlusion length is >1cm and ≤ 30 cm;
* Patient's reference vessel diameter is ≥ 4.0 mm and ≤6.0 mm (by visual angiographic estimation)
* Patient must be an acceptable candidate for PTA, peripheral artery bypass surgery or peripheral artery stent implantation;
* Female patients of child bearing potential must have a negative pregnancy test within 48 hours prior to the study procedure;
* Patient must have been informed of the nature of the study, agree to its provisions, and provide written informed consent;
* Patient is ≥ 21 years of age.

Exclusion Criteria:

* Patient has hypersensitivity or contraindication to aspirin, heparin, Plavix or radiographic contrast agents which cannot be adequately pre-medicated;
* The patient requires immediate treatment in more than one occluded vessel, in any combination of grafts or native vessels;
* Patient has planned femoropopliteal intervention scheduled within 30 days after index procedure;
* The patient is currently participating in another investigational drug or device trial that may conflict with study data collection and has not completed the entire follow-up period;
* Patient has no collateral flow distal to the occlusion;
* Patient's target occlusion has a dissection that occurred within the past 30 days caused by a guidewire attempt;
* Patient has a history of bleeding diatheses, coagulopathy or will refuse blood transfusion in cases of emergency;
* Patient suffered recent (within the past 6 months) significant gastrointestinal (GI) bleeding;
* Patient's target lesion or the vessel proximal to the target lesion reveals significant ectasia, dissection, aneurysm or thrombus;
* Patient has other medical illnesses (i.e., cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated with life-expectancy less than 1 year.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint of this study is to evaluate in hospital and 30 day major adverse events ("MAEs"), clinically significant perforations, clinically significant embolization and/or Grade C or greater dissections. | 30 days (+/-7 days)
Advancement of the ENABLER-P supported guidewire into or through the CTO in native femoropopliteal artery and subsequent achievement of distal vessel guidewire position with any conventional guidewire. | 30 days (+/-7 days)